CLINICAL TRIAL: NCT02073786
Title: : Rigid Video Stylet Can Provide More Successful Intubation Than Conventional Lightwand Intubation in Patients With Cervical Spine Operation : A Prospective Randomized Study
Brief Title: Rigid Video Stylet Vs Conventional Lightwand Intubation
Acronym: Optiscope
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Optiscope_SNUH
Record Dates: First submitted 2014-02-21; First posted 2014-02-27 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2014-02

CONDITIONS: Hoarseness; Intubation; Sorethroat
MeSH Terms: conditions — Hoarseness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lightwand (Active Comparator): Conventional lightwand intubation will performe for intubation
  Interventions: Device: Conventional lightwand intubation
- Optiscope (Experimental): Rigid video stylet, manufactural named Optiscope, will perform for intubation
  Interventions: Device: Rigid video stylet

INTERVENTIONS:
Device: Conventional lightwand intubation — Conventional lightwand intubation technique will perform during intubation
  Arms: Lightwand
Device: Rigid video stylet — Rigid video stylet will inserted through endotracheal tube before induction. After induction with propofol and remifentanil using TIVA infusion pump, rocuronium 0.6mg/kg were used to facilitate intubation. After 2minutes, board-certificated anesthesiologist perform intubation using Optiscope.
  Other Names: Optiscope® (Pacific Medical, Seoul, Republic of Korea)
  Arms: Optiscope

SUMMARY:
Lightwand is a useful alternative device for intubation but scooping movement can induce damage and microbleeding of oral mucosa, postoperative hoarseness,sore throat. Optiscope is rigid video stylet which has camera on distal tip of device. In many previous studies, rigid video stylet has proven advantages compared with other intubating devices.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for cervical spine surgery under general anesthesia
* aged between 20- 80 yrs

Exclusion Criteria:

* Patient who disagrees to participate this study
* Patient who has history of gastro-esophageal reflux disease, previous airway surgery, an increased risk of aspiration, coagulation disorders
* Patient who has congenital or acquired abnormalities of the upper airway, tumours, polyps, trauma, abscesses, inflammation or foreign bodies in the upper airway

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Primary success rate of intubation | within 90 sec from insertion of device
  compare primary success rate of intubation using Optiscope with lightwand intubation

SECONDARY OUTCOMES:
Intubation time | within 90 seconds from insertion of device
  Check the intubation time (sec) Intubation time defines "from insertion of device to oral cavity of patients to confirm successful intubation"
postoperative complications | During PACU stay time expected up to 1hr
  check the postoperative hoarseness, sorethroat and using numeric rating scale (0-10 point) we checked sorethroat score
postoperative complications | 24 hr after operation
  check the postoperative hoarseness, sorethroat and using numeric rating scale (0-10 point) we checked sorethroat score
hemodynamic change | baseline and 1minute after intubation
  check the changes of mean blood pressure, heart rate, pulse oximetry before and after intubation
number of intubation trial and scooping movements | during intubation time, an expected average of 1minute
  Check the number of intubation tiral and scooping movements during intubation

CONTACTS AND LOCATIONS:
Overall Officials: Hee Pyung Park, MD PhD, Study Director — Professor; Eugene Kim, MD, Principal Investigator — fellow
Locations (1):
- Seoul National University of Hospital, Seoul, South Korea